CLINICAL TRIAL: NCT07034118
Title: Definitive Proton Radiotherapy Combined With Chemotherapy and Immunotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma: A Phase I Clinical Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-ky212
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pronton radiotherapy with chemoimmunotherapy (Experimental): Pronton radiotherapy with chemoimmunotherapy
  Interventions: Radiation: Proton radiotherapy; Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Radiation: Proton radiotherapy — Patients enrolled would receive proton radiotherapy with chemoimmunotherapy.
Drug: Immune Checkpoint Inhibitors — Patients enrolled would receive proton radiotherapy and chemoimmunotherapy

SUMMARY:
The standard treatment for locally advanced esophageal squamous cell carcinoma (ESCC) is definitive concurrent chemoradiotherapy (CCRT). However, conventional photon-based radiotherapy is associated with excessive radiation exposure to normal tissues and a high incidence of treatment-related toxicities. Proton radiotherapy, one of the major advances in radiation oncology in recent years, offers the dosimetric advantage of reduced radiation to surrounding normal tissues, thereby decreasing the rate of adverse events. Two recent clinical studies have suggested that, compared with conventional photon radiotherapy, proton radiotherapy can significantly reduce the incidence of treatment-related toxicities and potentially improve patient survival outcomes.

Immune checkpoint inhibitors (ICIs) have been widely used in both locally advanced and advanced esophageal cancer and have demonstrated promising clinical efficacy. Preliminary results from several ongoing phase III clinical trials indicate that combining ICIs with concurrent chemoradiotherapy is both safe and effective. Moreover, proton radiotherapy, by minimizing the low-dose radiation exposure to circulating peripheral lymphocytes, may better preserve systemic immune function. Therefore, compared to photon therapy, proton radiotherapy may theoretically enhance the synergistic effect when combined with ICIs, offering a potential survival benefit.

Based on this rationale, we propose a phase I clinical trial to investigate the safety and preliminary efficacy of definitive proton chemoradiotherapy combined with immune checkpoint inhibition in patients with locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
1. Background Esophageal squamous cell carcinoma (ESCC) is a highly prevalent malignancy in China, ranking sixth in incidence and fourth in cancer-related mortality, posing a serious threat to public health. Over 50% of newly diagnosed patients present with locally advanced esophageal squamous cell carcinoma. The RTOG 8501 and RTOG 9405 trials established definitive concurrent chemoradiotherapy (CCRT) as the standard of care for inoperable locally advanced esophageal squamous cell carcinoma, yielding a 5-year overall survival (OS) rate of approximately 30%. However, despite optimization of physical radiation dose and fractionation in photon radiotherapy and modifications in chemotherapy regimens, further improvements in clinical outcomes have been limited.

   Recent research has focused on two primary strategies to enhance the efficacy of definitive CCRT in locally advanced esophageal squamous cell carcinoma: the incorporation of proton radiotherapy, and the integration of immune checkpoint inhibitors (ICIs).

   Conventional photon therapy using 6-8 MV X-rays typically involves a total dose of 50-60 Gy delivered over 28-30 fractions, with or without elective nodal irradiation (ENI). However, photon radiotherapy is limited by large gross tumor volumes (GTV) and widespread lymphatic involvement, leading to excessive radiation exposure to organs-at-risk (OARs). Elevated doses to the heart and lungs increase the risk of late toxicities such as radiation-induced heart disease and pulmonary fibrosis, thereby impairing cardiopulmonary function and survival. Additionally, high-dose exposure to circulating lymphocytes and the thoracic vertebrae compromises systemic immunity by inducing lymphopenia, adversely affecting prognosis.

   Proton radiotherapy, with its Bragg peak effect, delivers maximal radiation dose at the end of its range, significantly sparing surrounding normal tissues. Biologically, this translates into a lower incidence of late toxicities in the heart and lungs and reduced lymphocyte depletion, potentially leading to improved clinical outcomes. Emerging clinical data suggest that compared to conventional photon therapy, PRT reduces treatment-related toxicities and may improve survival.

   ICIs have shown promising efficacy in advanced EC and are increasingly being investigated in earlier disease stages. Several phase III trials (ESCORT-CRT, Keynote 975, RATIONAL 311, etc.) are evaluating the combination of CCRT with ICIs in locally advanced esophageal squamous cell carcinoma, and preliminary data indicate that this approach is both safe and effective. Since proton radiotherapy minimizes radiation dose to circulating lymphocytes, it may exhibit superior synergy with immunotherapy compared to photon radiotherapy, potentially offering enhanced therapeutic benefit.

   Therefore, we propose a Phase I clinical study to evaluate the safety and preliminary efficacy of definitive proton radiotherapy combined with chemotherapy and ICIs in patients with locally advanced esophageal squamous cell carcinoma.
2. Pretreatment Work-up

   1. Physical exam and ECOG assessment
   2. PET-CT or contrast-enhanced CT of neck, chest, and abdomen (PET-CT preferred) to confirm staging
   3. Upper GI endoscopy and esophagography
   4. Peripheral blood sample collection
   5. Tumor biopsy sample acquisition for pathological confirmation
3. Proton Radiotherapy Protocol 3.1 Simulation

   1. Large-bore CT simulator with IV contrast; slice thickness ≤5 mm
   2. Immobilization using thermoplastic mask or vacuum cushion 3.2 Target Delineation Involved-field irradiation (IFI) plus elective nodal irradiation (ENI) GTV: primary tumor and involved lymph nodes CTV: GTV + 3 cm cranio-caudal and 0.8 cm radial margins; include involved nodal stations

ENI regions per JES classification:

Cervical: bilateral 101, 102, 104, 105, 106rec Upper thoracic: bilateral 101, 104, 105, 106, part of 108 Middle thoracic: bilateral 101, 104, 105, 106, 107, 108, partial 110, abdominal groups 1, 2, 3, 7 Lower thoracic: 107, 108, 110, abdominal groups 1, 2, 3, 7 PTV: CTV + 6 mm margin Prescribed dose: 50.4 GyE in 28 fractions 3.3 Dosimetric Planning

1. Pencil beam scanning with multi-field optimization (MFO)
2. Field arrangement: 2 oblique beams for upper EC; 2-3 oblique fields form middle/lower EC
3. Setup: 5 mm field margin, 3.5% range uncertainty
4. Dose constraints: PTV: 100% covered by 95% of prescribed dose; Lungs: V20 <23%, V5 <50%, Dmean <13 GyE; Spinal cord: Dmax <45 GyE; Heart: V40 <10%, Dmean 15-20 GyE; Liver: V20 <33%, Dmean <13 GyE; Kidneys: V20 <20%, Dmean <13 GyE 3.4 Treatment Delivery Daily image guidance using CBCT. After 10 fractions, tumor response assessed; if significant shrinkage, re-simulation and field adaptation required 3.5 Pharmacologic Therapy Concurrent chemotherapy: Nab-paclitaxel 125 mg/m² on days 1 and 8, Carboplatin AUC = 5 on day 1 Concurrent immunotherapy: Immune checkpoint inhibitor on day 1, every 3 weeks, for 2 cycles Post-radiotherapy: If no grade ≥3 adverse events, maintenance immunotherapy every 3 weeks for up to 1 year 3.6 Follow-Up Schedule

During Radiotherapy:

Weekly: CBC, liver/kidney function, stool routine/occult blood After 10 fractions: Weekly esophagography After 23 fractions: Contrast-enhanced CT of neck, chest, abdomen

Post-Radiotherapy (4 weeks):

Chest CT to assess for acute radiation pneumonitis Every 3 months: Contrast-enhanced CT (neck/chest/abdomen), esophagography During immunotherapy maintenance: Monthly labs including cardiac enzymes, myoglobin, thyroid and adrenal function, SCC antigen

After Completion of Immunotherapy:

Years 1-3: CT and esophagography every 3 months, gastroscopy annually Years 4-5: CT and esophagography every 6 months, gastroscopy annually After year 5: Annual CT, esophagography, and gastroscopy

ELIGIBILITY:
Inclusion Criteria:

Age 18-75 years ECOG performance status 0-1 Histologically confirmed esophageal squamous cell carcinoma (ESCC) Stage II-IVA disease (AJCC 8th edition), confirmed via contrast-enhanced CT of the neck, chest, and abdomen, or PET-CT Unresectable by surgical evaluation or patient refusal of surgery No prior oncologic treatment Life expectancy >6 months Radiotherapy plan meets physical dose constraints Signed informed consent by patient or legal representative

Exclusion Criteria:

Age <18 or >75 years ECOG >1 or inability to tolerate treatment Histology other than squamous cell carcinoma Stage I or IVB disease High risk of hemorrhage or fistula, as assessed by imaging and radiation oncologists Previously treated patients Life expectancy <6 months Contraindications to chemotherapy or immunotherapy Radiotherapy plan fails to meet dose constraints Lack of signed informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity | One year
  The incidence of myelosuppression, radiation-induced pneumonitis and esophagitis, radiation-induecd cardiac injury, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No